CLINICAL TRIAL: NCT06805253
Title: Left Ventricular Reverse Remodeling Outcomes Evaluation in Patients With Aortic Regurgitation After Surgical Treatment
Brief Title: Left Ventricular Reverse Remodeling Evaluation After Surgical Correction of Aortic Regurgitation
Acronym: ORMIX
Status: Recruiting | Type: Observational
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Collaborators: Voronezh regional clinical hospital #1 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 173538086
Record Dates: First submitted 2024-10-18; First posted 2025-02-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Regurgitation; Mitral Valve Regurgitation; Left Ventricle Dilated; Left Atrium Dilated; Systolic Left Ventricular Heart Failure; Diastolic Heart Failure
Keywords: reverse remodeling; left ventricle dilatation; mitral valve functional regurgitation recovery; left ventricle reverse remodeling
MeSH Terms: conditions — Aortic Valve Insufficiency; Mitral Valve Insufficiency; Heart Failure, Diastolic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MR < 2 no MvR: Patients with functional mitral regurgitation grade 0-1, 1 and 1-2 without mitral valve repair (MvR)
  Interventions: Other: Not applicable - observational study
- MR >= 2 no MvR: Patients with mitral valve functional regurgitation of grade 2 and more severe without mitral valve repair
  Interventions: Other: Not applicable - observational study
- MR < 2 MvR: Patients with functional mitral regurgitation grade 0-1, 1 and 1-2, mitral valve repaired
  Interventions: Other: Not applicable - observational study
- MR >= 2 MvR: Patients with mitral valve functional regurgitation of grade 2 and more severe, mitral valve repaired
  Interventions: Other: Not applicable - observational study

INTERVENTIONS:
Other: Not applicable - observational study — observation only
  Other Names: observation

SUMMARY:
Investigators assume that surgical correction approach to functional mitral regurgitation during intervention for chronic aortic regurgitation in patients with severe enlargement of the left heart chambers influences reverse remodeling of the left ventricle (LV) in the postoperative period. It is suggested that functional mitral regurgitation (MR) provides supra-physiological left ventricle volume overload and this fact plays positive role in early-stage post-operative left ventricle volume and function recovery. LV volume, systolic and diastolic function will be monitored with echocardiography (EchoCG) along with life quality in patients with different grades of functional mitral regurgitation secondary to severe chronic aortic insufficiency after surgical treatment of aortic regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Planned primary elective surgery for chronic aortic regurgitation
* Presence of functional mitral regurgitation
* End-diastolic volume of the left ventricle >= 250 ml

Exclusion Criteria:

* Infectious endocarditis
* History of myocardial infarction
* Indications on simultaneous myocardial revascularisation
* Acute aortic regurgitation of any etiology
* Previously diagnosed dilatation of the left ventricle, not associated with the development of aortic regurgitation
* Long-term persistent or permanent form of atrial fibrillation
* Pregnancy in the first 12 months after surgery
* Simultaneous participation in other studies
* Presence of implanted pacemakers
* Refusal to sign informed consent
* Acute coronary event diagnosed within 12 months after aortic valve surgery
* Indications for resynchronization therapy or permanent right ventricular pacing in the first 12 months after aortic valve surgery
* Re-do cardiac surgery for any reason within 12 months after aortic valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent open surgical correction of aortic insufficiency with the background of severe eccentric remodeling of the left ventricle (EDV more than 250 ml). Men and women over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
LV end-diastolic volume (EDV) decrease | 3 and 12 months after surgery
  Change in end-diastolic volume of the left ventricle, assessed with EchoCG after surgical correction of aortic insufficiency
Freedom from readmission | 12 months after surgery
  Freedom from readmission due to valvular problem or heart failure-related reason

SECONDARY OUTCOMES:
Life quality | Upon inclusion, 10 days post-surgery, 3 month and 12 month post-surgery
  The patient's life quality according to the results of the EuroQol-5D-5L (EQ-5D-5L) questionnaire (0-100 points, the higher - the better).

OTHER OUTCOMES:
LV ejection fraction (EF) | 3 and 12 month post-surgery
  Left ventricle ejection fraction, assessed with EchoCG
LV diastolic function | Upon inclusion, 3 month and 12 month post-surgery
  Left ventricle diastolic function, assessed with EchoCG
Left atrium volume index (LAVI) | Upon inclusion, 3 month and 12 month post-surgery
  Left atrium volume indexed to body surface area, assessed with EchoCG

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Petrovsky National Research Center of Surgery, Moscow
  - Voronezh Regional Clinical Hospital No. 1, Voronezh

DOCUMENTS (1):
  • Study Protocol (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT06805253/Prot_000.pdf